CLINICAL TRIAL: NCT05928585
Title: Phase 1 Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HIB210 in Healthy Volunteers
Brief Title: A Study of Safety and Drug Levels of HIB210 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HI-Bio, A Biogen Company (Industry)
Responsible Party: Sponsor
Organization: Biogen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIB-210-101
Record Dates: First submitted 2023-06-12; First posted 2023-07-03 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Immune System Diseases; Autoimmunity
Keywords: C5aR1; C5a receptor; C5aR1 inhibition; CD88
MeSH Terms: conditions — Immune System Diseases; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAD HIB210 (Experimental): Increasing doses of HIB210 will be administered for cohorts 1-4 in a multiple ascending dose format
  Interventions: Drug: HIB210
- MAD Placebo (Placebo Comparator): Placebo will be administered for cohorts 1-4 in a multiple ascending dose format
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HIB210 — Experimental monoclonal antibody
  Arms: MAD HIB210
Drug: Placebo — Placebo
  Arms: MAD Placebo

SUMMARY:
The goal of this clinical trial is to test safety of the investigational product in healthy volunteers. The main questions it aims to answer is when HIB210 is administered as multiple doses, is it:

1. Safe
2. Well tolerated
3. Does the body absorb and eliminate HIB210 as expected

DETAILED DESCRIPTION:
Study Sponsor, originally HI-Bio, Inc., is now HI-Bio, A Biogen Company.

ELIGIBILITY:
Key Eligibility Criteria:

* Healthy male and females between 19 to 65 years of age
* Normal or not significantly abnormal laboratory tests and EKG findings during Screening
* No significant medical conditions that might affect ability to participate in the study or present a safety risk
* No evidence of significant or recurrent infection or recent infection
* No history of cancer other than certain skin cancers and limited cancer of the cervix of the womb
* Willingness to comply with birth control requirements of the study (for both men and women)
* No recent major surgery or trauma or planned surgery during the study or within 1 month after the study
* Body mass index (BMI) between 18 and 32 kg/m2

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Baseline to End of Study (Up to Day 114)
Number of participants with clinical laboratory abnormalities | Baseline to End of Study (Up to Day 114)
Number of participants with electrocardiogram (ECG) abnormalities | Baseline to End of Study (Up to Day 114)
Number of participants with physical examination abnormalities | Baseline to End of Study (Up to Day 114)
Number of participants with vital sign abnormalities | Baseline to End of Study (Up to Day 114)

SECONDARY OUTCOMES:
PK Parameters: Cmax | Baseline to Day 29
  Maximum Serum Concentration (Cmax)
PK Parameters: tmax | Baseline to Day 29
  Time to Maximum Serum Concentration (tmax)
PK Parameters: AUC | Baseline to Day 29
  Area under the serum concentration-time curve
Anti-drug Antibodies (ADA) | Baseline to End of Study (Up to Day 114)
  Baseline prevalence and post-dose incidence of ADA

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — HI-Bio, A Biogen Company
Locations (1):
- HI-Bio Investigational Site, Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/